CLINICAL TRIAL: NCT02469337
Title: Randomized Control Trial of Dichloroacetate, Preoperative Carbohydrate Loading and Moderate Intensity Exercise on Muscle Insulin Resistance After Major Abdominal Surgery
Brief Title: Role of Preoperative Carbohydrates Drinks, Dichloroacetate and Exercise on Postoperative Muscle Insulin Resistance
Acronym: CARBEX
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 11/EE/0395
Record Dates: First submitted 2015-06-08; First posted 2015-06-11 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Dichloroacetic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Preoperative carbohydrate drinks (Active Comparator): Patients who were randomised to carbohydrate group ingested 800ml PreOp (Nutricia Clinical Care, 12.5g CHO/100 ml) the night before and 400ml in the morning of surgery, about 2-3 hours before the induction of anaesthesia.
  Interventions: Dietary Supplement: Carbohydrate drinks
- Dichloroacetate infusion (Active Comparator): The patients in the dichloroacetate group received the CHO drinks as well as an intravenous infusion of DCA (50mg/kg body weight) over 45 min, one- two hours before the induction of anaesthesia.
  Interventions: Drug: Dichloroacetate
- Moderate intensity exercise (Active Comparator): Patients randomised to exercise group, will perform a 30 min exercise using a semi-recumbent exercise bike, at about 70% of their age estimated heart rate(determined by the formula: (220-Age)*0.7 under close supervision and monitoring of their vital parameters.
  Interventions: Behavioral: Moderate intensity exercise
- Control (No Intervention): Patients in this group will have surgery as standard practice with none of the above interventions

INTERVENTIONS:
Drug: Dichloroacetate — Dichloroacetate, an analog of acetic acid has been shown to increase the activation of PDC by inhibiting PDK4 in humans. This drug is expected to shift the metabolism of pyruvate from glycolysis and towards oxidative pathway in the mitochondria
  Other Names: sodium dichloroacetate
  Arms: Dichloroacetate infusion
Dietary Supplement: Carbohydrate drinks — preoperative carbohydrate drinks
  Arms: Preoperative carbohydrate drinks
Behavioral: Moderate intensity exercise — 30 min exercise using a semi-recumbent exercise bike, at about 70% of their age estimated heart rate
  Arms: Moderate intensity exercise

SUMMARY:
The aim of the study is to investigate whether preoperative interventions such as carbohydrate drinks, Dichloroacetate and exercise would inhibit or reverse the changes in molecular mechanisms regulating muscle carbohydrate oxidation and postoperative muscle insulin resistance in patients undergoing major abdominal surgery.

DETAILED DESCRIPTION:
Forty patients undergoing open elective gastrointestinal surgery, will be randomized to four groups of 10 each. The patients will be randomised to receive either preoperative (1) oral carbohydrate drinks (CHO) or (2) infusion of Dichloroacetate with oral carbohydrate drinks (3) exercise or (4) standard care.

Since the interventions are qualitatively different and only the physiological mechanisms are being studied rather than the clinical outcomes, the study is not blinded and no placebo is used.

Analysis for cytokines, insulin, glucagon levels will be performed at screening, during surgery and on the 2nd postoperative day. Muscle biopsies will be taken at the beginning and end of surgery, from rectus abdominus and vastus lateralis muscles for analysis of mRNA (IL-6, TNF-α, Akt1, IRS-1, FOXO1, MAFbx, MURF1 and PDK4) and protein (MafBx, FOXO1, PDK4) expression and muscle metabolites (glycogen, lactate, triglycerides and FFA). Oral Glucose Tolerance Test (GTT) to be performed at the screening visit and on the 2nd postoperative day using a standard protocol. The techniques to be employed to study the above will include RT-PCR, radioimmunoassay, spectophotometry, bioluminometry, Western blotting and ELISA.

Primary outcome: The changes in indices of muscle insulin resistance and muscle protein breakdown at the beginning and at the end of surgery, in response to surgical stress.

Secondary outcomes: (a) The expression of muscle metabolites, reflecting muscle protein turnover (b) Clinical Outcomes: Length of stay and incidence of postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 years of age, who are undergoing major elective open abdominal surgery will be included in the study. Patients should be able to provide a written informed consent to participate in the study.

Exclusion Criteria:

* Patients who are

  1. Undergoing emergency surgery
  2. Suffering from chronic illness, (e.g. diabetes) or other debilitating diseases
  3. On long term anti-inflammatory drugs, (e.g. NSAIDS, Steroids, immunosuppressant)
  4. On long term antibiotics
  5. On Statins
  6. On full therapeutic dose of anticoagulants, or aspirin >325 mg/day, Clopidrogel >75mg/day
  7. Suffering from bleeding diathesis
  8. Unable to give consent
  9. Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-05; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
insulin resistance | 48 hours after surgery
  Relative changes in indices of muscle insulin resistance namely PDC activity, PDK4 mRNA and protein expression.

SECONDARY OUTCOMES:
muscle carbohydrate oxidation | 48 hours after surgery
  Changes in muscle metabolites such as glycogen, glucose, lactate, reflecting the changes in skeletal muscle carbohydrate oxidation.
Mitochondrial ATP production | 48 hours after surgery
  Mitochondrial ATP production rates in patients undergoing major abdominal surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Dileep N Lobo, Professor, Principal Investigator — University of Nottingham
Locations (1):
- University Hospitals Nottingham Queen's Medical Centre, Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No